CLINICAL TRIAL: NCT05423470
Title: Effect of Intermittent Hypoxia on Ischemia-reperfusion Injury in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sophie Lalande, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018110129
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Intermittent Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent hypoxia (Experimental): The intermittent hypoxia protocol will consist of three 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with 4-minute normoxic cycles.
  Interventions: Behavioral: Intermittent hypoxia
- Intermittent normoxia (Sham Comparator): The intermittent normoxia protocol will consist of three 4-minute normoxic cycles (compressed air) interspersed with 4-minute normoxic cycles (room air).
  Interventions: Behavioral: Intermittent normoxia

INTERVENTIONS:
Behavioral: Intermittent hypoxia — The intermittent hypoxia protocol will consist of three 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with 4-minute normoxic cycles.
  Arms: Intermittent hypoxia
Behavioral: Intermittent normoxia — The intermittent normoxia protocol will consist of three 4-minute normoxic cycles (compressed air) interspersed with 4-minute normoxic cycles (room air).
  Arms: Intermittent normoxia

SUMMARY:
The objective of the present study is to determine whether intermittent hypoxia protects against ischemia-reperfusion injury in young and older healthy individuals. The investigators hypothesize that intermittent hypoxia will attenuate the reduction in flow-mediated dilation following ischemia-reperfusion injury.

DETAILED DESCRIPTION:
Ischemic heart disease represents the most common form of cardiovascular disease and the main cause of mortality in the United States. Ischemic heart disease originates from an inadequate blood supply to the coronary arteries. While immediate reperfusion of the tissues represents the first-line treatment for ischemia, restoration of blood flow causes further damage to the endothelial cells lining the blood vessels. Indeed, severe endothelial dysfunction occurs paradoxically during the initial period of reperfusion, partly due to oxidative stress caused by a burst of reactive oxygen species formation and a reduction in nitric oxide bioavailability. Ischemia-reperfusion injury represents the endothelial damage caused by the combined effects of ischemia and reperfusion. Myocardial ischemia-reperfusion injury induces coronary endothelial dysfunction, which in turn promotes myocardial infarction. Thus, interventions designed to attenuate the effect of ischemia-reperfusion injury are urgently needed to prevent myocardial injury in patients with ischemic heart disease.

The endothelial function of the brachial artery strongly correlates with coronary artery endothelial function. Accordingly, measures of brachial artery function such as flow-mediated dilation can act as a surrogate of coronary artery endothelial function. Flow-mediated dilation, an indicator of nitric oxide-dependent endothelial function, represents the dilation of the brachial artery following increases in blood flow and shear stress induced by a transient period of ischemia. A standard model of ischemia-reperfusion injury consists of occluding blood flow to the arm for a period of 20 minutes. This prolonged forearm occlusion causes a reduction in flow-mediated dilation ranging from 30 to 50% for at least 30 minutes after reperfusion in young individuals.

Local ischemic preconditioning offers protection against ischemia-reperfusion injury. Ischemic preconditioning consists of exposing an individual to repeated brief periods of ischemia, induced by inflating a cuff on the upper arm, before an ischemia-reperfusion injury. Ischemic preconditioning (3 cycles of 5-minute ischemia followed by 5 minutes of reperfusion) applied immediately before ischemia-reperfusion injury prevents the reduction in flow-mediated dilation in healthy individuals, suggesting that ischemic preconditioning could be protective in patients with acute ischemia about to undergo therapeutic reperfusion. The protection provided by ischemic preconditioning appears to depend on the activation of adenosine triphosphate-sensitive potassium channel. Therefore, ischemic preconditioning attenuates the impaired endothelial-dependent dilation from subsequent, prolonged ischemia-reperfusion injury in humans.

Intermittent hypoxia represents a potential systemic strategy to prevent the reduction in flow-mediated dilation following ischemia-reperfusion injury. Intermittently breathing mildly hypoxic air stimulates an endothelium-dependent dilation and prevents endothelial dysfunction through the production of reactive oxygen species and an increase in nitric oxide bioavailability. Short periods of intermittent hypoxia in animal models induces ischemic preconditioning and protect the heart from subsequent infarction. Indeed, intermittent hypoxia conditioning consisting of 5-8 cycles/day for 5-10 min/cycle at a fraction of inspired oxygen of 9.5-10% interspersed with 4 min normoxia over a period of 20 days protected the endothelium-dependent dilation of coronary and systemic arteries in rats through activation of free-radical processes. Moreover, intermittent hypoxia consisting of 5 cycles of 6-minutes of hypoxia at an oxygen concentration of 6% interspersed with 6 minutes of exposure to room air over 1 hour significantly reduced infarct size in hearts from mice when performed 24 hours before ischemia-reperfusion injury, in association with hypoxia-inducible factor expression. Intermittent hypoxia may therefore induce protection via a systemic response representing a distinct mechanism from the local protective response induced by brief ischemic preconditioning.

Healthy aging results in a greater decrease in flow-mediated dilation following blood flow occlusion. Indeed, decreases in flow-mediated dilation ranging from 50 to 68% were observed in middle-aged men, due to further oxidative stress and reduced nitric oxide bioavailability. While ischemic preconditioning prevented the decrease in flow-mediated dilation in young healthy individuals, the preventive effect of ischemic preconditioning against ischemia-reperfusion injury was abolished in older individuals. However, ischemic preconditioning significantly attenuated the decrease in flow-mediated dilation in older patients with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years old

Exclusion Criteria:

* Have high blood pressure (above 130/80 mmHg)
* Are smokers
* Are pregnant
* Have a history of cardiovascular disease, diabetes or lung disease
* Are taking medication affecting the cardiovascular system
* Carpal tunnel syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in endothelial-dependent vasodilation of the brachial artery will be assessed by flow-mediated dilation using an ultrasound machine | Measured before and 15 minutes after an ischemia-reperfusion injury.
  Indicator of nitric oxide-dependent endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lalande, Principal Investigator — UT Austin
Locations (1):
- The Unviersity of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kvietys PR, Granger DN. Endothelial cell monolayers as a tool for studying microvascular pathophysiology. Am J Physiol. 1997 Dec;273(6):G1189-99. doi: 10.1152/ajpgi.1997.273.6.G1189. PMID 9435543
- [Background] Csiszar A, Wang M, Lakatta EG, Ungvari Z. Inflammation and endothelial dysfunction during aging: role of NF-kappaB. J Appl Physiol (1985). 2008 Oct;105(4):1333-41. doi: 10.1152/japplphysiol.90470.2008. Epub 2008 Jul 3. PMID 18599677
- [Background] Grisham MB, Granger DN, Lefer DJ. Modulation of leukocyte-endothelial interactions by reactive metabolites of oxygen and nitrogen: relevance to ischemic heart disease. Free Radic Biol Med. 1998 Sep;25(4-5):404-33. doi: 10.1016/s0891-5849(98)00094-x. PMID 9741579
- [Background] Honda HM, Korge P, Weiss JN. Mitochondria and ischemia/reperfusion injury. Ann N Y Acad Sci. 2005 Jun;1047:248-58. doi: 10.1196/annals.1341.022. PMID 16093501
- [Background] Powers SK, Murlasits Z, Wu M, Kavazis AN. Ischemia-reperfusion-induced cardiac injury: a brief review. Med Sci Sports Exerc. 2007 Sep;39(9):1529-36. doi: 10.1249/mss.0b013e3180d099c1. PMID 17805085
- [Background] Rodriguez-Manas L, El-Assar M, Vallejo S, Lopez-Doriga P, Solis J, Petidier R, Montes M, Nevado J, Castro M, Gomez-Guerrero C, Peiro C, Sanchez-Ferrer CF. Endothelial dysfunction in aged humans is related with oxidative stress and vascular inflammation. Aging Cell. 2009 Jun;8(3):226-38. doi: 10.1111/j.1474-9726.2009.00466.x. Epub 2009 Feb 26. PMID 19245678
- [Background] Anderson TJ, Uehata A, Gerhard MD, Meredith IT, Knab S, Delagrange D, Lieberman EH, Ganz P, Creager MA, Yeung AC, et al. Close relation of endothelial function in the human coronary and peripheral circulations. J Am Coll Cardiol. 1995 Nov 1;26(5):1235-41. doi: 10.1016/0735-1097(95)00327-4. PMID 7594037
- [Background] Harris RA, Nishiyama SK, Wray DW, Richardson RS. Ultrasound assessment of flow-mediated dilation. Hypertension. 2010 May;55(5):1075-85. doi: 10.1161/HYPERTENSIONAHA.110.150821. Epub 2010 Mar 29. PMID 20351340
- [Background] Aboo Bakkar Z, Fulford J, Gates PE, Jackman SR, Jones AM, Bond B, Bowtell JL. Prolonged forearm ischemia attenuates endothelium-dependent vasodilatation and plasma nitric oxide metabolites in overweight middle-aged men. Eur J Appl Physiol. 2018 Aug;118(8):1565-1572. doi: 10.1007/s00421-018-3886-z. Epub 2018 May 21. PMID 29785503
- [Background] Brunt VE, Jeckell AT, Ely BR, Howard MJ, Thijssen DH, Minson CT. Acute hot water immersion is protective against impaired vascular function following forearm ischemia-reperfusion in young healthy humans. Am J Physiol Regul Integr Comp Physiol. 2016 Dec 1;311(6):R1060-R1067. doi: 10.1152/ajpregu.00301.2016. Epub 2016 Oct 5. PMID 27707723
- [Background] Devan AE, Umpierre D, Harrison ML, Lin HF, Tarumi T, Renzi CP, Dhindsa M, Hunter SD, Tanaka H. Endothelial ischemia-reperfusion injury in humans: association with age and habitual exercise. Am J Physiol Heart Circ Physiol. 2011 Mar;300(3):H813-9. doi: 10.1152/ajpheart.00845.2010. Epub 2011 Jan 14. PMID 21239631
- [Background] DeVan AE, Umpierre D, Lin HF, Harrison ML, Tarumi T, Dhindsa M, Hunter SD, Sommerlad SM, Tanaka H. Habitual resistance exercise and endothelial ischemia-reperfusion injury in young adults. Atherosclerosis. 2011 Nov;219(1):191-3. doi: 10.1016/j.atherosclerosis.2011.07.099. Epub 2011 Jul 26. PMID 21840524
- [Background] Loukogeorgakis SP, Williams R, Panagiotidou AT, Kolvekar SK, Donald A, Cole TJ, Yellon DM, Deanfield JE, MacAllister RJ. Transient limb ischemia induces remote preconditioning and remote postconditioning in humans by a K(ATP)-channel dependent mechanism. Circulation. 2007 Sep 18;116(12):1386-95. doi: 10.1161/CIRCULATIONAHA.106.653782. Epub 2007 Aug 27. PMID 17724264
- [Background] Carden DL, Granger DN. Pathophysiology of ischaemia-reperfusion injury. J Pathol. 2000 Feb;190(3):255-66. doi: 10.1002/(SICI)1096-9896(200002)190:33.0.CO;2-6. PMID 10685060
- [Background] Gross GJ, Auchampach JA. Blockade of ATP-sensitive potassium channels prevents myocardial preconditioning in dogs. Circ Res. 1992 Feb;70(2):223-33. doi: 10.1161/01.res.70.2.223. PMID 1310443
- [Background] Chang HR, Lien CF, Jeng JR, Hsieh JC, Chang CW, Lin JH, Yang KT. Intermittent Hypoxia Inhibits Na+-H+ Exchange-Mediated Acid Extrusion Via Intracellular Na+ Accumulation in Cardiomyocytes. Cell Physiol Biochem. 2018;46(3):1252-1262. doi: 10.1159/000489076. Epub 2018 Apr 16. PMID 29672298
- [Background] Mateika JH, El-Chami M, Shaheen D, Ivers B. Intermittent hypoxia: a low-risk research tool with therapeutic value in humans. J Appl Physiol (1985). 2015 Mar 1;118(5):520-32. doi: 10.1152/japplphysiol.00564.2014. Epub 2014 Dec 30. PMID 25549763
- [Background] Manukhina EB, Belkina LM, Terekhina OL, Abramochkin DV, Smirnova EA, Budanova OP, Mallet RT, Downey HF. Normobaric, intermittent hypoxia conditioning is cardio- and vasoprotective in rats. Exp Biol Med (Maywood). 2013 Dec;238(12):1413-20. doi: 10.1177/1535370213508718. Epub 2013 Nov 4. PMID 24189016
- [Background] Cai Z, Manalo DJ, Wei G, Rodriguez ER, Fox-Talbot K, Lu H, Zweier JL, Semenza GL. Hearts from rodents exposed to intermittent hypoxia or erythropoietin are protected against ischemia-reperfusion injury. Circulation. 2003 Jul 8;108(1):79-85. doi: 10.1161/01.CIR.0000078635.89229.8A. Epub 2003 Jun 9. PMID 12796124
- [Background] van den Munckhof I, Riksen N, Seeger JP, Schreuder TH, Borm GF, Eijsvogels TM, Hopman MT, Rongen GA, Thijssen DH. Aging attenuates the protective effect of ischemic preconditioning against endothelial ischemia-reperfusion injury in humans. Am J Physiol Heart Circ Physiol. 2013 Jun 15;304(12):H1727-32. doi: 10.1152/ajpheart.00054.2013. Epub 2013 Apr 19. PMID 23604707
- [Background] Burtscher M, Haider T, Domej W, Linser T, Gatterer H, Faulhaber M, Pocecco E, Ehrenburg I, Tkatchuk E, Koch R, Bernardi L. Intermittent hypoxia increases exercise tolerance in patients at risk for or with mild COPD. Respir Physiol Neurobiol. 2009 Jan 1;165(1):97-103. doi: 10.1016/j.resp.2008.10.012. Epub 2008 Nov 1. PMID 19013544
- [Background] Burtscher M, Pachinger O, Ehrenbourg I, Mitterbauer G, Faulhaber M, Puhringer R, Tkatchouk E. Intermittent hypoxia increases exercise tolerance in elderly men with and without coronary artery disease. Int J Cardiol. 2004 Aug;96(2):247-54. doi: 10.1016/j.ijcard.2003.07.021. PMID 15262041
- [Background] Wesseling KH, Jansen JR, Settels JJ, Schreuder JJ. Computation of aortic flow from pressure in humans using a nonlinear, three-element model. J Appl Physiol (1985). 1993 May;74(5):2566-73. doi: 10.1152/jappl.1993.74.5.2566. PMID 8335593
- [Background] Seeger JP, Benda NM, Riksen NP, van Dijk AP, Bellersen L, Hopman MT, Cable NT, Thijssen DH. Heart failure is associated with exaggerated endothelial ischaemia-reperfusion injury and attenuated effect of ischaemic preconditioning. Eur J Prev Cardiol. 2016 Jan;23(1):33-40. doi: 10.1177/2047487314558377. Epub 2014 Nov 11. PMID 25389072
- [Background] Laurie SS, Yang X, Elliott JE, Beasley KM, Lovering AT. Hypoxia-induced intrapulmonary arteriovenous shunting at rest in healthy humans. J Appl Physiol (1985). 2010 Oct;109(4):1072-9. doi: 10.1152/japplphysiol.00150.2010. Epub 2010 Aug 5. PMID 20689088